CLINICAL TRIAL: NCT07172932
Title: ANTIBIOTIC-RESISTANT ENTEROBACTERALES BLOODSTREAM INFECTIONS AND RISK FACTORS IN PATIENTS ADMITTED TO THE INTENSIVE CARE UNIT
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Fahriye Melis Gürsoy Kurtoğlu, specialist doctor, Ankara City Hospital Bilkent
Other Study IDs: E1-21-2215
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Bloodstream Infections; Enterobacteriaceae Infections; Intensive Care (ICU); Antibiotic Resistant Infection
Keywords: Bloodstream Infections; esbl; carbapenem resistance; colistin resistance
MeSH Terms: conditions — Sepsis; Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we first aimed to reveal the resistance profile of Enterobacteriales bloodstream infections at our center.

We evaluated data from patients with ESBL, colistin, and carbapenem resistance and identified resistance risk factors.

We then reviewed our approach to managing the infection based on the results obtained.Patients were grouped according to resistance patterns and resistance status and compared retrospectively.

DETAILED DESCRIPTION:
Antibiotic resistance represents one of the most urgent and serious challenges confronting modern healthcare systems. This problem is particularly critical in intensive care units (ICUs), where bloodstream infections (BSIs) caused by resistant organisms are frequently associated with prolonged hospitalization, increased healthcare costs, therapeutic failures, and high mortality rates.

Over the past decade, the incidence of bloodstream infections due to Enterobacterales species has risen substantially worldwide. These pathogens possess diverse resistance mechanisms that undermine the effectiveness of commonly used antibiotics. Among the most clinically significant are extended-spectrum beta-lactamases (ESBLs), carbapenemase production, and the emergence of colistin resistance phenotypes. These mechanisms not only limit empiric treatment options but also complicate infection control practices and contribute to the spread of multidrug-resistant organisms across healthcare facilities.

In Turkey, national and multicenter surveillance data indicate that resistance rates among ICU isolates of Klebsiella pneumoniae and Escherichia coli often exceed the European average. This situation directly impacts empiric antibiotic therapy by reducing the likelihood of initial treatment success, while also facilitating the nosocomial transmission of resistant strains. Consequently, optimizing empiric therapy strategies and strengthening infection control measures are of paramount importance in ICUs.

The present study was designed to retrospectively evaluate all cases of Enterobacterales bloodstream infections (EBSIs) diagnosed in our center between 2019 and 2022. The primary objectives were:

To identify the prevalence and distribution of key antibiotic resistance phenotypes (including ESBL, carbapenem, and colistin resistance).

To analyze patient- and treatment-related risk factors associated with the emergence of resistance.

To assess the potential clinical consequences of resistance in terms of morbidity, mortality, and therapeutic outcomes.

To provide evidence-based data that may inform and support the development of local infection control policies and antimicrobial stewardship interventions.

By systematically examining the resistance patterns and associated risk factors in a large cohort of ICU patients, this study aims to contribute to a better understanding of the epidemiology of resistant Enterobacterales infections. Furthermore, the findings are expected to provide valuable insights for revising empiric treatment guidelines and for guiding infection control strategies tailored to high-risk patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Isolation of an Enterobacterales species from a blood culture obtained during ICU stay
* The isolate considered as the causative pathogen by an Infectious Diseases and Clinical Microbiology specialist

Exclusion Criteria:

* Isolates not considered as causative pathogens
* Growth of a different pathogen in blood culture within ±72 hours of the index culture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study included adult patients who were hospitalized in the intensive care units (ICUs) of the Neurology-Orthopedics Building at Ankara City Hospital between September 2019 and December 2022. Eligible participants were aged 18 years or older and had a blood culture positive for Enterobacterales species during ICU stay, which was evaluated by an Infectious Diseases and Clinical Microbiology specialist as the causative pathogen.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of antibiotic resistance phenotypes (ESBL, carbapenem, colistin) among Enterobacterales bloodstream infection isolates. | From January 2019 to December 2022
  Prevalence of antibiotic resistance phenotypes (ESBL, carbapenem, colistin) among Enterobacterales bloodstream infection isolates.

SECONDARY OUTCOMES:
Identification of patient-related and clinical risk factors associated with antibiotic-resistant Enterobacterales bloodstream infections. | 2019-2022.
  Risk factors such as age, comorbidities, prior antibiotic use, invasive device utilization (mechanical ventilation, central venous catheter, urinary catheter), and ICU stay will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No